CLINICAL TRIAL: NCT06657014
Title: Caregiver Mind-Mindedness Training as an Early Intervention for Reducing Social Anxiety in Preschool-Aged Children: A Randomized Controlled Trial
Brief Title: Caregiver Mind-Mindedness Training to Alleviate Social Anxiety in Children
Acronym: CAMPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heriot-Watt University (Other)
Responsible Party: Principal Investigator, Hiva Javadian, Doctoral Researcher, Heriot-Watt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-SOCIALANXIETY-2024; Heriot watt university (Other: Heriot watt university)
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Social Anxiety Disorder of Childhood
Keywords: Mind-Mindedness; Social Anxiety; intervention

STUDY DESIGN:
Intervention Model Description: The Mind-Mindedness Training group will participate in three structured online sessions aimed at enhancing caregivers' ability to recognize and respond to their child's thoughts and feelings. This training seeks to improve caregivers' mentalization, which may help reduce social anxiety symptoms in children. Meanwhile, the Peer Support group will have access to a private online platform where caregivers can share experiences and coping strategies, creating a supportive environment without the structured intervention.
  Data will be collected at baseline, immediately after the intervention, and during a three-month follow-up to assess changes in mind-mindedness, child social anxiety, attachment styles, and theory of mind. This parallel assignment model enables an effective evaluation of the intervention's impact on the target population while controlling for external variables through random assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-Mindedness Training Group (Experimental): The Mind-Mindedness Training Group will involve 50 caregivers of preschool-aged children (ages 4 to 7) with social anxiety. Participants will attend three one-hour online sessions over three consecutive weeks.
  The training focuses on enhancing caregivers' ability to recognize and respond to their children's thoughts and emotions. Each session includes:
  * Session 1:** Introduction to mind-mindedness, its importance, and caregiver roles in managing social anxiety.
  * Session 2:** Practical strategies for emotion coaching, including role-play exercises.
  * Session 3:** Advanced strategies addressing common challenges, with discussions and video examples.
  Participants will receive materials to support their learning. Effectiveness will be assessed through evaluations of mind-mindedness, child social anxiety, and related areas at baseline, post-intervention, and three months later.
  Interventions: Other: mind-mindedness
- Peer Support Control Group (Active Comparator): The Peer Support Control Group will consist of 50 primary caregivers of preschool-aged children (ages 4 to 7) exhibiting signs of social anxiety. Participants will not receive Mind-Mindedness training but will have access to a private online peer support platform.
  This group aims to provide a supportive environment for caregivers to share experiences, concerns, and coping strategies. Key features include:
  Peer Support Platform:A moderated online group for discussions and emotional support among caregivers.
  Resource Sharing: Opportunities for caregivers to share helpful articles, tips, and resources.
  Facilitated Discussions: Occasional prompts to encourage conversations about common challenges.
  Participants will complete assessments of mind-mindedness, social anxiety, attachment, and theory of mind at baseline, post-intervention, and three months later, similar to the Mind-Mindedness Training Group. This control group allows for comparisons of the effectiveness
  Interventions: Other: mind-mindedness

INTERVENTIONS:
Other: mind-mindedness — The Mind-Mindedness Training Intervention is a structured program designed specifically for primary caregivers of preschool-aged children (ages 4 to 7) who exhibit signs of social anxiety. This intervention is unique because it focuses on enhancing caregivers' understanding and responsiveness to their children's emotional and mental states through the concept of mind-mindedness.

SUMMARY:
This randomized controlled trial (RCT) aims to investigate the efficacy of Mind-Mindedness (MM) training for caregivers as an early intervention for preschool-aged children (4 to 7 years) exhibiting signs of social anxiety. The study posits that enhancing caregivers' ability to recognize and respond to their children's thoughts, feelings, and intentions-termed Mind-Mindedness-can foster secure attachments and improve socioemotional outcomes for children.

A total of 100 primary caregivers will be recruited from the United Kingdom and Iran, with participants randomly assigned to either an MM training intervention group or a peer support control group. The MM training will consist of three online sessions, each lasting one hour, focusing on strategies for implementing mind-minded comments and enhancing emotional understanding. The peer support group will provide caregivers with an online platform for sharing experiences related to their child's anxiety without receiving structured training.

Assessments of Mind-Mindedness, child social anxiety, attachment, and theory of mind will be conducted at baseline, post-intervention, and three months after the intervention using validated measures. This study aims to evaluate the effectiveness of MM training in reducing social anxiety symptoms in children while examining the potential mediating roles of attachment and theory of mind in this relationship.

By incorporating a cross-cultural approach, this research will contribute to understanding the influence of cultural contexts on the effectiveness of caregiver interventions. The anticipated findings could establish MM training as a valuable strategy for mitigating social anxiety in preschoolers and inform future clinical practices aimed at enhancing caregiver-child interactions.

DETAILED DESCRIPTION:
This study aims to explore a new approach to support preschool children (ages 4 to 7) who struggle with social anxiety. The investigators believe that when caregivers, such as parents, understand and respond more effectively to their child's feelings and thoughts, it can help the child feel more secure and less anxious in social situations.

To test this idea, the investigators are inviting 100 caregivers from the UK and Iran to participate in our research. Participants will be randomly divided into two groups: one group will receive special training called Mind-Mindedness training, which consists of three online sessions designed to teach caregivers techniques for better understanding their child's emotions. The other group will participate in a peer support group where participants can share experiences with other caregivers, this group will not receive the training.

The investigators will assess the children's social anxiety before the training, immediately after it, and three months later to determine if the training has a positive impact. This study aims to demonstrate how enhancing caregiver awareness of their child's feelings can reduce anxiety and help children interact more confidently with others.

ELIGIBILITY:
Inclusion Criteria:

* Primary Caregiver Status: Participants must be the primary caregiver of a child aged 4 to 7 years.

Age of Caregiver: Caregivers must be between 18 and 60 years old. Geographical Location: Caregivers must reside in either the United Kingdom or Iran.

Social Anxiety Symptoms: Children must exhibit observable signs of social anxiety, which will be confirmed through a standardized screening tool.

Exclusion Criteria:

* Clinical Diagnosis: Children with a clinical diagnosis of another psychiatric disorder (e.g., autism spectrum disorder, ADHD) will be excluded.

Concurrent Support: Caregivers of children who are currently receiving any other form of psychological support or treatment for social anxiety will be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Child Social Anxiety Levels | Data will be collected at baseline, immediately after the intervention, and at a 3-month follow-up
  Primary Outcome Measure
  Description: This measure will assess changes in social anxiety symptoms in preschool-aged children (4 to 7 years) as reported by caregivers, using the Spence Children's Anxiety Scale (SCAS), the parent versions. The SCAS scores range from a minimum of 0 to a maximum of 114. Higher scores on the SCAS indicate worse outcomes, reflecting higher levels of anxiety.

SECONDARY OUTCOMES:
Mind-Mindedness of Caregivers | Data will be collected at baseline, immediately after the intervention, and at a 3-month follow-up.
  The assessment of mind-mindedness in caregivers will be conducted using the Mind-Mindedness Coding Manual(Meins, 2015). It evaluates caregivers' ability to understand and respond to their child's mental and emotional states. Scores on this scale typically range from 0 to 5, with higher scores indicating better outcomes, reflecting a greater level of mind-mindedness. A higher score signifies that the caregiver is more attuned to their child's emotional needs, which is associated with positive developmental outcomes for the child.

OTHER OUTCOMES:
Attachment Security of Children | Data will be collected at baseline, immediately after the intervention, and at a 3-month follow-up.
  The assessment of attachment in caregivers will be conducted using the Attachment Insecurity Screening Inventory (AISI), developed by Spruit et al. (2018), allowing the evaluation of any changes in attachment security resulting from the intervention. This scale has a scoring range from 0 to 30, with higher scores indicating worse outcomes and greater attachment insecurity. Therefore, a higher score suggests that the caregiver exhibits more insecure attachment behaviours.
Theory of Mind Development in Children | Data will be collected at baseline, immediately after the intervention, and at a 3-month follow-up.
  The Theory of Mind Task Battery (Hutchins et al., 2012) will be utilized to assess children's understanding of others' mental states, an important factor in social interactions and emotional regulation. Scores on this battery typically range from 0 to 30, with higher scores indicating better outcomes. A higher score reflects a greater ability for the child to understand and interpret the mental states of others, which is crucial for social interactions and emotional development.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hale, Asst. Prof., Study Director — Herriot Watt University
Locations (1):
- Heriot watt, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers for several reasons:
  1. Participant Privacy: Protecting the privacy and confidentiality of participants is our highest priority. Sharing IPD could compromise their anonymity.
  2. Data Sensitivity: The data collected during the trial may contain sensitive information that requires strict confidentiality measures.
  3. Ethical Considerations: Ethical guidelines related to participant consent prohibit sharing identifiable data without explicit permission.

REFERENCES:
- [Derived] Javadian H, Stewart ME, Mathews M, Williams AJ, Hale D. Caregiver mind-mindedness training as an early intervention for social anxiety in children: A protocol for a randomised controlled trial. PLoS One. 2025 Sep 22;20(9):e0315150. doi: 10.1371/journal.pone.0315150. eCollection 2025. PMID 40982456